CLINICAL TRIAL: NCT04087655
Title: NADPH Oxidase Activity and Muscle Microvascular Dysfunction in Obesity
Brief Title: Microvascular Dysfunction in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Bob Hickner, Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R15HL113854 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2019-09-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Endothelial Dysfunction
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single group of obese adults studied before and after exercise training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Experimental): Eight weeks of interval exercise training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Eight weeks of interval exercise training

SUMMARY:
Impaired endothelial function is observed in disease states related to obesity, such as atherosclerosis, coronary artery disease, and diabetes. Reactive oxygen species (ROS) production and resultant oxidative stress contribute to the development of these obesity-related diseases. The enzyme NADPH-oxidase is a major source of oxidative stress within the vasculature, and has been linked with the Metabolic Syndrome. In the investigator's previously funded studies, the investigators demonstrated for the first time that: 1) in vivo ROS were elevated in skeletal muscle of obese as compared to lean or overweight human subjects, 2) perfusion of the NADPH-oxidase inhibitor apocynin locally into muscle normalized ROS levels and reversed local microvascular endothelial dysfunction in the obese individuals, and 3) aerobic exercise training was effective at attenuating in vivo hydrogen peroxide production and reversing microvascular endothelial dysfunction in the obese individuals. The investigators will investigate in this R15 renewal application the mechanism of exercise training-induced alterations in ROS production and action on endothelial dysfunction in obesity using our newly developed microdialysis methodology of monitoring ROS production, in combination with analysis of muscle biopsy samples obtained before and after our previously tested 8-week intervention of aerobic interval exercise training. The objectives of this study are to determine the impact of in vivo NADPH oxidase activity on endothelial function in obese individuals, and to determine the mechanism of training-induced improvements in endothelial function. The investigator's unique microdialysis methodology will allow monitoring of microvascular/endothelial function and ROS generation, as well as the administration of pharmacological agents directly into muscle. The central hypothesis is that it is upregulation of both mitochondrial ROS and NADPH oxidase-derived ROS that results in endothelial dysfunction in obesity, and that exercise training down-regulates mitochondrial-derived ROS, and NADPH oxidase 4, thereby improving endothelial function. The aims of this proposal are to: 1) determine the contributions of mitochondrial ROS and specific NADPH oxidase isoforms to the NADPH oxidase dependent endothelial dysfunction in skeletal muscle of obese individuals; 2) determine the mechanism of ROS reduction and improved endothelial function resulting from an 8-week aerobic interval training program.

DETAILED DESCRIPTION:
Twenty-five sedentary class 2 and above obese [body mass index (BMI) >35 kg/m2, waist circumference >40 inches (men) or >35 inches (women)] men and women (18-45 yrs) will participate in these experiments. Individuals under 18 years of age will not be investigated due to the invasive nature of the protocol. Individuals greater than 45 years of age will not be investigated due to the age-related decline in endothelial function. There will be no restrictions with regard to race, sex, or socioeconomic status. Women will be premenopausal, will be on combined estrogen/progestin hormonal contraceptive therapy (oral pill, transdermal patch or vaginal ring) and will be studied within the seven day inactive (placebo) phase of hormonal contraceptive therapy (comparable to the early follicular phase in the normal menstrual cycle; verified by blood estradiol analyses). Ensuring consistency in studying the women during the phase of hormonal contraceptive therapy with lowest plasma estradiol concentrations is important due to the known positive effects of estradiol on endothelial function. Sedentary obese individuals will have been weight stable for the preceding 6 months, and will have the Metabolic Syndrome. The Metabolic Syndrome will be defined according to the most widely used criteria for the Metabolic Syndrome from the Third Report of the National Cholesterol Education Program Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Individuals with the Metabolic Syndrome have at least three of the following:1) Central obesity as measured by waist circumference (men >40 inches; women >35 inches); 2) Fasting blood triglycerides > 150 mg/dL; 3) Blood HDL cholesterol in men<40 mg/dL and women <50 mg/dL; 4) Blood pressure > 130/85 mmHg; 5) Fasting blood glucose > 110 mg/dL, and (not per ATP III) a 2-hour GTT glucose of 140-200 mg/dl.

Before participating in this study, subjects will undergo a medical history, physical examination, and screening for cardiovascular disease and type 2 diabetes. Evaluations consist of a graded treadmill stress test, a blood chemistry, body composition analysis by Dual X-ray Absorptiometry (DXA) and a minimum waist circumference (between the xiphoid process and the umbilicus) measure.

Exclusions Subjects participating in purposeful endurance exercise training (>20 min/day, >1 day/week) will be excluded. Pre-menopausal female subjects must not be pregnant or lactating, and must have had regular menstrual cycles for the past year. All subjects will be screened for cardiovascular and peripheral vascular disease. Individuals taking medications that may affect central or peripheral circulation, are on nonsteroidal anti-inflammatory agents or serotonin reuptake inhibitors, who smoke or chew tobacco, have diabetes (fasting blood glucose >125 mg/dL), hypertension >160/95 mmHg (individuals with diabetes and high degree of hypertension will be excluded to keep a more uniform group of individuals with the metabolic syndrome), congestive heart failure, angina, or peripheral vascular disease. Individuals with evidence of serious arrhythmias and/or acute myocardial ischemia reflected in ST-segment depression of 1 mm or greater at rest or during exercise will be excluded. Individuals with chronic infections, paralysis due to stroke, advanced Parkinson's Disease, severe rheumatoid arthritis or other serious orthopedic problems that would prevent performance of the exercise training tasks will be excluded. Subjects will not be allowed to take antioxidant, herbal or vitamin supplementation for at least 2 weeks prior to investigation since some of these agents have been shown to improve endothelium-dependent vasodilatation. Subjects will not be allowed to ingest caffeine the day of the experiment. Subjects will be excluded if weight changes by more than 5% during the training program or if their exercise adherence is below 90% of the exercise sessions or total exercise time.

Timeframe: Subjects will be recruited, screened, enrolled, and tested during months 3-28 of this grant. Subject recruitment procedures and procurement of needed supplies will occur during the first 2 months of the project. Additional recruitment, as well as screening and testing of subjects will occur in 1-month cycles over the ensuing 25 months at a rate of approximately 1 per cycle. Twenty-five microdialysis experiments will therefore be performed on participants both before and after 8 weeks of exercise training, for a total of 50 microdialysis experiments. This plan will therefore require 2 microdialysis tests per month on average during the testing months. Testing of these subjects includes six hours for the microdialysis procedure. Biochemical analysis of samples requires approximately six hours per experiment, and data reduction another five hours per experiment. Additional time (five hours per week) is required for subject recruitment, preliminary testing and follow-up. The recruitment and testing goals are therefore realistic in light of the personnel and percentage efforts allocated, coupled with personnel and resources not charged to the grant.

Microdialysis (Before and after exercise training):

Subjects will report to the Hickner laboratory following an overnight fast. While subjects are quietly resting, an overnight fasted blood draw will be obtained from an antecubital vein to be analyzed for traditional (insulin, glucose, lipids, c-reactive protein) and non-traditional [(cytokines TNF-alpha, IL-6, IL-13, intercellular adhesion molecule-1 (ICAM-1), vascular adhesion molecule-1 (VCAM-1) and P-selectin] cardio-metabolic disease risk/inflammatory markers in blood using ELISA's from EMD Millipore, or our clinical analyzer (Beckman Access systems). In addition, plasma glutathione (GSH/GSSG) will be analyzed as a marker of systemic oxidative stress using a kit from Percipio Biosciences (Bioxytech GSH/GSSG).

Microdialysis Procedure Seven microdialysis probes (CMA 20: 10mm * 0.5 mm 20kilodalton cutoff membrane, 5 cm probe shaft length, inlet tubing and outlet tubing 20cm; CMA/Microdialysis, Stockholm, Sweden) will be percutaneously inserted, 3 cm apart, into the vastus lateralis of the quadriceps femoris muscle group (3-4 probes per leg) using sterile technique under local anesthesia (1% lidocaine). The probes will be perfused with the appropriate solution at a rate of 2.0 µL/min using CMA/102 microinfusion pumps (CMA/Microdialysis, Stockholm, Sweden) according to the schedule in Table 2.

The control perfusion solution will consist of a sterile saline solution containing 5 mM ethanol (for blood flow/microvascular exchange measures). Two of the probes will initially be perfused with this control solution while the other probes will be perfused with NADPH oxidase inhibitors. Subjects will rest while seated for 60 minutes to allow for recovery from probe insertion and equilibration of the perfusate with the local environment. Phase 1: Three 10-minute dialysate samples will be collected over the subsequent 30 minutes in capped 150 µL polyethylene collection vials to determine basal nutritive flow in the absence (probe 1) and presence (Probes 3-7) of the NADPH oxidase inhibitors, and to serve as an intra-probe control period prior to SNP perfusion (Probe 2). Phase 2: The perfusate solutions in the second probe will then be changed to contain the control solution plus 50 mM sodium nitroprusside (SNP: to control for non-endothelium dependent changes). 100 µM Amplex UltraRed and 1 U/mL horseradish peroxidase (HRP) will be added to the perfusate in the other probes for measurement of in vivo H2O2 production. Three twenty-minute dialysate samples will then be collected over the subsequent 60 minutes to provide these measures in the absence of superoxide dismutase. Phase 3: 10 U/mL superoxide dismutase (SOD) will then be added to the Amplex UltraRed/HRP containing perfusates. Three twenty-minute dialysate samples will then be collected over the subsequent 60 minutes to provide measures of the effects of SNP, 1 mM apocynin, 100nM MitoTempo,100uM MitoTempo+Apocynin, 100nM GKT 137831, or 100nM GKT 137831+Apocynin in the absence of SOD. Phase 4: The perfusate solutions in probes two through seven will then be changed to contain the control solution plus either 50 mM Ach (to determine endothelium-dependent changes), or 50 mM ACh + either 1 mM apocynin, 100nM MitoTempo,100uM MitoTempo+Apocynin, 100nM GKT 137831, or 100nM GKT 137831+Apocynin (to determine if inhibition of NADPH oxidase or mitochondrial ROS production improves the endothelium-dependent response). The probes will then be perfused for 60 minutes to allow for equilibration with the local environment. Three ten-minute samples will then be collected over the subsequent 30 minutes to determine the nutritive flow effects of ACH in the presence and absence of NADPH oxidase or mitochondrial ROS inhibition. For each sample where Amplex UltraRed and HRP are added to the perfusion medium, 30 µL of dialysate will immediately be measured for H2O2 in the laboratory fluorometer. For each sample where blood flow is measured, dialysate will be stored at 4 °C and analyzed for ethanol (for blood flow/microvascular exchange) within 24 hours. All perfusates and dialysates will be protected from light exposure.

Microdialysis ethanol outflow/inflow ratio Ethanol (5 mM) will be included in the perfusion medium to monitor nutritive blood flow/microvascular exchange in the area of the microdialysis probe as described in our previous publications 30-32.

Determination of peak aerobic capacity (before and after exercise training):

All subjects will perform a standardized maximal exercise test on a treadmill upon enrollment in the study and again upon completion of the training program. Subjects will individually adjust speed and incline (3-6 km·hr-1, 0-5%) for a 5-minute warm-up period. After the warm-up period, the subject's expired O2 and CO2 will be continuously monitored via open circuit spirometry (TrueOne 2400; Parvomedics; Salt Lake City, UT). The VO2peak test will be performed using a ramp protocol where the speed will be constant and the incline will be increased 2% every two-minutes until VO2peak is reached. The starting speed will be individually adjusted based on the warm-up speeds and heart rates, with the intention of obtaining VO2peak within 8-12 minutes.

Training Protocol All participants will perform aerobic interval exercise training three times per week on non-consecutive days for eight weeks. Exercise will consist of walking/running up an incline on a treadmill. Subjects will warm up for 10 minutes at 70% of maximal heart rate (HRmax as determined during the VO2peak test) before performing four 4-minute intervals at 90% of HRmax with a 3-minute active recovery at 70% of HRmax between intervals and a 5-minute cool-down period, yielding a total exercise time of 40 minutes.

Determination of body composition Fat-free mass, fat mass, and percent body fat will be determined using dual-energy x-ray absorptiometry (DXA; GE Lunar Prodigy Advance, Madison WI). Body mass and height will be measured for the calculation of body mass index (BMI: kg/m2). Minimum waist and maximum hip circumferences will be also measured to potentially be used as a covariate in statistical analyses due to the relationship of w/h ratio and waist circumference with cardio-metabolic disease risk.

Muscle markers of oxidative stress:

Biopsies will therefore be taken in the resting state before and after training in those participants agreeing to the biopsy procedure. Percutaneous muscle biopsies will be obtained from the vastus lateralis of the quadriceps femoris muscle group (undergoes adaptations to the proposed exercise training) using sterile procedures and after administration of local anesthesia (1% lidocaine).

ELIGIBILITY:
Inclusion Criteria:

* There will be no restrictions with regard to race, sex, or socioeconomic status.
* Women will be premenopausal
* Women will be on combined estrogen/progestin hormonal contraceptive therapy (oral pill, transdermal patch or vaginal ring).
* Sedentary obese individuals will have been weight stable for the preceding 6 months.
* Sedentary obese individuals will have the Metabolic Syndrome as defined according to the Third Report of the National Cholesterol Education Program Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III).
* Individuals with the Metabolic Syndrome will have at least three of the following:

  1. Central obesity as measured by waist circumference (men >40 inches; women >35 inches);
  2. Fasting blood triglycerides > 150 mg/dL;
  3. Blood HDL cholesterol in men<40 mg/dL and women <50 mg/dL;
  4. Blood pressure > 130/85 mmHg; 5) Fasting blood glucose > 110 mg/dL, and (not per ATP III) a 2-hour GTT glucose of 140-200 mg/dl.

Exclusion Criteria:

* Subjects participating in purposeful endurance exercise training (>20 min/day, >1 day/week) will be excluded.
* Pre-menopausal female subjects must not be pregnant or lactating, and must have had regular menstrual cycles for the past year.
* Individuals taking medications that may affect central or peripheral circulation,
* Individuals on nonsteroidal anti-inflammatory agents or serotonin reuptake inhibitors,
* Individuals who smoke or chew tobacco,
* Individuals with diabetes (fasting blood glucose >125 mg/dL),
* hypertension >160/95 mmHg
* Individuals with congestive heart failure, angina, or peripheral vascular disease. --Individuals with ECG evidence of serious arrhythmias and/or acute myocardial ischemia reflected in ST-segment depression of 1 mm or greater at rest or during exercise.
* Individuals with chronic infections, paralysis due to stroke, advanced Parkinson's Disease, severe rheumatoid arthritis or other serious orthopedic problems that would prevent performance of the exercise training tasks will be excluded.
* Individuals taking antioxidant, herbal or vitamin supplementation for at least 2 weeks prior to investigation.
* Individuals ingesting caffeine the day of the experiment.
* Individuals whose weight changes by more than 5% during the training program.
* Individuals whose exercise adherence is below 90% of the exercise sessions or total exercise time.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Reactive oxygen species (ROS) | change from week 0 to week 8
  reactive oxygen species as indicated by H2O2 concentration measured with microdialysis

SECONDARY OUTCOMES:
Muscle blood flow | change from week 0 to week 8
  muscle microvascular blood flow as monitored with microdialysis

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Hickner, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04087655/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04087655/SAP_001.pdf